CLINICAL TRIAL: NCT00385450
Title: Cardiopulmonary Bypass-Induced Lymphocytopenia and the Potential Effects of Protease Inhibitor in the Perioperative Period
Brief Title: Cardiopulmonary Bypass-Induced Lymphocytopenia and the Potential Effects of Protease Inhibitor
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study closed at Mayo prior to completion
Sponsor: Mayo Clinic (Other)
Responsible Party: IRBe Secretary-Ben Wibstad, IRBe
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: 05-004052 00
Record Dates: First submitted 2006-10-05; First posted 2006-10-09 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2015-04

CONDITIONS: Cardiopulmonary Bypass
MeSH Terms: interventions — Nelfinavir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nelfinavir/placebo (Experimental)
  Interventions: Drug: Nelfinavir/placebo

INTERVENTIONS:
Drug: Nelfinavir/placebo — 1250mg/twice each day/four days.

SUMMARY:
In previous studies, 90% of patients who underwent elective cardiopulmonary bypass procedure manifested CD4 counts of less than 500 cells/microliter in the immediate (day 1) post-operative period. This study will investigate whether or not Nelfinavir increases those CD4 counts in the post-operative period.

DETAILED DESCRIPTION:
See Brief Summary.

ELIGIBILITY:
Inclusion Criteria:

* Any patient undergoing elective (non-emergency) cardiopulmonary bypass for coronary artery bypass grafting, cardiac valve replacement, or both.

Exclusion Criteria:

* A dozen different medical conditions and two dozen medical contraindications.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2006-10; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Proportion of Nelfinavir patients v. proportion of placebo patients who have CD4 counts of less than 500 cells/microliter | Six days.

SECONDARY OUTCOMES:
Changes in quantitative measure of inflammatory markers | Six days.
Changes in clinical outcomes. | Six days.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew D. Badley, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States